CLINICAL TRIAL: NCT02948829
Title: An Open Label, Phase 2 Study to Investigate Cell-mediated Immunity and Safety of a Tetravalent Dengue Vaccine Candidate (TDV) Administered Subcutaneously in Healthy Children Aged 4 to 16 Years
Brief Title: Safety and Immunogenicity of Takeda's Tetravalent Dengue Vaccine (TDV) in Healthy Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DEN-313; U1111-1184-1893 (Other: WHO)
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tetravalent Dengue Vaccine (TDV) 0.5 mL (Experimental): TDV 0.5 mL, subcutaneous (SC) injection, on Day 1 (Month 0) and Day 90 (Month 3).
  Interventions: Biological: TDV

INTERVENTIONS:
Biological: TDV — TDV SC injection.

SUMMARY:
The purpose of this study is to assess the cellular immune responses following 2 doses given 3 months apart of tetravalent dengue vaccine candidate (TDV) in 4 to 16 years' healthy participants.

DETAILED DESCRIPTION:
The vaccine tested in this study was TDV. This study assessed cellular immune responses and safety up to 3 years post second TDV administration to healthy children aged 4 to 16 years and in dengue endemic regions.

The study enrolled 200 participants. Participants received:

• TDV 0.5 mL subcutaneous (SC) injection into the upper arm at Day 1 (Month 0) and at Day 90 (Month 3).

This multi-center trial was conducted in Panama and Philippines. 198 participants received the 2-dose schedule of TDV, and 2 participants received only the first dose of TDV (Day 1). Participants made multiple visits to the clinic and were contacted at least every week for the entire study duration post first injection.

ELIGIBILITY:
Main Inclusion Criteria:

1. Is aged 4 to 16 years, inclusive (Latin America) or 4 to 8 years, inclusive (Asia).
2. Are in good health at the time of entry into the study as determined by medical history, physical examination (including vital signs), and clinical judgment of the investigator.

Main Exclusion Criteria:

1. Febrile illness (body temperature ≥38°C) or moderate or severe acute illness or infection at the time of enrolment.
2. History or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose an additional risk to the participant due to participation in the study.
3. Receipt of any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to Day 1 (Month 0) or planning to receive any vaccines within 28 days after Day 1 (Month 0).
4. Previous participation in any clinical study of a dengue candidate vaccine, or previous receipt of any dengue vaccines (investigational or licensed).

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- CEVAXIN, Panama City, Panama
- Research Institute for Tropical Medicine, City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Panama and Philippines from 03 April 2017 to 14 December 2020.
Pre-assignment Details: Healthy participants were enrolled in a single arm in this study to receive 2 doses of Tetravalent Dengue Vaccine (TDV) injection subcutaneously (SC).
Period: Overall Study
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Started | 200
Completed | 184
Not Completed | 16
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject and/or Subject's Parent(s)/ Legally Authorized Representative (LAR) | 5
Not completed — Pregnancy | 1
Not completed — Other: Reason not Specified | 8

BASELINE CHARACTERISTICS:
Population: Safety Set included all enrolled participants who received at least 1 dose of TDV.
Groups:
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3).
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.7 (2.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 76
  Asian | 100
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 9
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Panama | 100
  Philippines | 100
Height [Mean (Standard Deviation); unit: cm] | 118.38 (14.564)
Weight [Mean (Standard Deviation); unit: kg] | 23.54 (10.258)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = weight (kg)/[height (m)^2]
  kg/m^2 | 16.15 (3.104)
Baseline Seropositivity Status [Count of Participants; unit: Participants] — Seropositive at Baseline was defined as a reciprocal neutralizing titer >=10 for one or more dengue serotypes. Seronegative at Baseline was defined as having a reciprocal neutralizing titer <10 for all dengue serotypes. The 4 dengue virus serotypes were dengue virus (DENV)-1, DENV-2, DENV-3 and DENV-4.
  Participants
    Seropositive | 113
    Seronegative | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cellular Immune Response to 2 Doses of Tetravalent Dengue Vaccine (TDV) at 1 Month Post Second Vaccination
Description: Percentage of participants with cellular immune response were reported. Cellular immune response was defined as an interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) response that was >3 times higher compared to Baseline (Day 1) and ≥ 5 spots per well. Cellular immune response to any peptide pool was reported. The peptide pool included non-structural proteins (NS) NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2. Percentage of participants with cellular immune response were reported. Percentages are rounded off to the nearest decimal point.
Time Frame: 1 month post second vaccination (Day 120)
Population: Per-Protocol Set (PPS) included all participants from the Full Analysis Set (FAS) who have no major protocol violations. Overall number of participants analyzed are participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 173
percentage of participants | 97.1 [93.4 to 99.1]

2. Secondary Outcome: Magnitude of Cellular Immune Response Assessed by Number of Spot Forming Cells (SFC)/Million Peripheral Blood Mononuclear Cells (PBMCs) Measured by IFN-γ ELISPOT at 1 Month Post Second Vaccination
Description: The magnitude of cellular immune response was assessed by the number of SFC/million PBMCs for participants with a cellular immune response. Cellular immune response was defined as IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1) and ≥ 5 spots per well. Data (SFC/million PBMC) for participants with a cellular immune response to any peptide pool is reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2.
Time Frame: 1 month post second vaccination (Day 120)
Population: PPS included all participants from the FAS who have no major protocol violations. Overall number of participants analyzed are participants with data available for analysis.
Measure: Median (Inter-Quartile Range); unit: SFC/million PBMCs
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 168
SFC/million PBMCs | 846.5 [378.5 to 1968.5]

3. Secondary Outcome: Percentage of Participants With Cellular Immune Response to TDV at 1 Month Post First Vaccination, Pre-second Vaccination, 6 Months Post Second Vaccination, and Annually at Years 1, 2, and 3
Description: Percentage of participants with cellular immune response were reported. Cellular immune response was defined as an IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1 [M0]) and >=5 spots per well. Cellular immune response to any peptide pool was reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2. Percentages are rounded off to the nearest decimal point.
Time Frame: 1 month post first vaccination (Day 30); pre-second vaccination (Day 90); 6 months post second vaccination (Day 270); Years 1, 2 and 3
Population: PPS included all participants from the FAS who have no major protocol violations. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 195
percentage of participants
  Day 30: number analyzed (Participants) | 171
  Day 30 | 95.3 [91.0 to 98.0]
  Day 90: number analyzed (Participants) | 183
  Day 90 | 95.1 [90.9 to 97.7]
  Day 270: number analyzed (Participants) | 173
  Day 270 | 95.4 [91.1 to 98.0]
  Year 1: number analyzed (Participants) | 174
  Year 1 | 90.8 [85.5 to 94.7]
  Year 2: number analyzed (Participants) | 150
  Year 2 | 84.0 [77.1 to 89.5]
  Year 3: number analyzed (Participants) | 171
  Year 3 | 77.8 [70.8 to 83.8]

4. Secondary Outcome: Magnitude of Cellular Immune Response Assessed by Number of SFC/Million PBMCs Measured by IFN-γ ELISPOT at 1 Month Post First Vaccination, Pre-second Vaccination, 6 Months Post Second Vaccination, and Annually at Years 1, 2, and 3
Description: as for outcome 2
Time Frame: 1 month post first vaccination (Day 30); pre-second vaccination (Day 90); 6 months post second vaccination (Days 120 and 270); Years 1, 2 and 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: SFC/million PBMCs
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 195
SFC/million PBMCs
  Day 30: number analyzed (Participants) | 163
  Day 30 | 1019.0 [418.0 to 2542.0]
  Day 90: number analyzed (Participants) | 174
  Day 90 | 536.5 [254.0 to 1212.0]
  Day 270: number analyzed (Participants) | 165
  Day 270 | 486.0 [203.0 to 1252.0]
  Year 1: number analyzed (Participants) | 158
  Year 1 | 193.0 [76.0 to 482.0]
  Year 2: number analyzed (Participants) | 126
  Year 2 | 104.0 [41.0 to 560.0]
  Year 3: number analyzed (Participants) | 133
  Year 3 | 136.0 [47.0 to 577.0]

5. Secondary Outcome: Percentage of Participants With Cellular Immune Responses to TDV at 1 Month Post First Vaccination, Pre-second Vaccination, 1 and 6 Months Post Second Vaccination, and Annually at Years 1, 2, and 3 Assessed by Country
Description: Percentage of participants with cellular immune response by country were reported. Cellular immune response was defined as an IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1 [M0]) and >=5 spots per well. Cellular immune response to any peptide pool was reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2. Data is reported as per enrollment by country (Panama and Philippines). Percentages are rounded off to the nearest decimal point.
Time Frame: 1 month post first vaccination (Day 30); pre-second vaccination (Day 90) 1 and 6 months post second vaccination (Days 120 and 270); Years 1, 2, 3
Population: PPS 'by country' included all participants from the FAS who have no major protocol violations. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: Panama: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants from Panama.
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: Philippines: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants from Philippines.
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Panama | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Philippines
Number analyzed (Participants) | 97 | 98
percentage of participants
  Day 30: number analyzed (Participants) | 76 | 95
  Day 30 | 96.1 [88.9 to 99.2] | 94.7 [88.1 to 98.3]
  Day 90: number analyzed (Participants) | 85 | 98
  Day 90 | 96.5 [90.0 to 99.3] | 93.9 [87.1 to 97.7]
  Day 120: number analyzed (Participants) | 75 | 98
  Day 120 | 97.3 [90.7 to 99.7] | 96.9 [91.3 to 99.4]
  Day 270: number analyzed (Participants) | 75 | 98
  Day 270 | 94.7 [86.9 to 98.5] | 95.9 [89.9 to 98.9]
  Year 1: number analyzed (Participants) | 83 | 91
  Year 1 | 91.6 [83.4 to 96.5] | 90.1 [82.1 to 95.4]
  Year 2: number analyzed (Participants) | 52 | 98
  Year 2 | 86.5 [74.2 to 94.4] | 82.7 [73.7 to 89.6]
  Year 3: number analyzed (Participants) | 79 | 92
  Year 3 | 79.7 [69.2 to 88.0] | 76.1 [66.1 to 84.4]

6. Secondary Outcome: Percentage of Participants With Cellular Immune Responses to TDV:1 Month Post First Vaccination, Pre-second Vaccination, 1 and 6 Months Post Second Vaccination, and Annually at Years 1, 2, and 3, by Dengue Baseline Seropositivity Status
Description: Percentage of participants with cellular immune response by dengue Baseline seropositivity status were reported. Cellular immune response was defined as an IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1 [M0]) and >=5 spots per well. Seropositive at Baseline was defined as a reciprocal neutralizing titer >=10 for one or more dengue serotypes. Seronegative at Baseline was defined as having a reciprocal neutralizing titer <10 for all dengue serotypes. The 4 dengue virus serotypes were dengue virus (DENV)-1, DENV-2, DENV-3 and DENV-4. Cellular immune response to any peptide pool was reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2. Data is reported per Baseline seropositivity status of participants (Seropositive and Seronegative). Percentages are rounded off to the nearest decimal point.
Time Frame: 1 month post first vaccination (Day 30); pre-second vaccination (Day 90); 1 and 6 months post second vaccination (Days 120 and 270); Years 1, 2, and 3
Population: PPS 'by Baseline seropositivity status' included all participants from the FAS who have no major protocol violations. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: Seropositive: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants seropositive at Baseline.
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: Seronegative: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants seronegative status at Baseline.
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Seropositive | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Seronegative
Number analyzed (Participants) | 109 | 86
percentage of participants
  Day 30: number analyzed (Participants) | 97 | 74
  Day 30 | 91.8 [84.4 to 96.4] | 100.0 [95.1 to 100.0]
  Day 90: number analyzed (Participants) | 104 | 79
  Day 90 | 93.3 [86.6 to 97.3] | 97.5 [91.2 to 99.7]
  Day 120: number analyzed (Participants) | 100 | 73
  Day 120 | 96.0 [90.1 to 98.9] | 98.6 [92.6 to 100.0]
  Day 270: number analyzed (Participants) | 101 | 72
  Day 270 | 93.1 [86.2 to 97.2] | 98.6 [92.5 to 100.0]
  Year 1: number analyzed (Participants) | 98 | 76
  Year 1 | 87.8 [79.6 to 93.5] | 94.7 [87.1 to 98.5]
  Year 2: number analyzed (Participants) | 93 | 57
  Year 2 | 80.6 [71.1 to 88.1] | 89.5 [78.5 to 96.0]
  Year 3: number analyzed (Participants) | 97 | 74
  Year 3 | 74.2 [64.3 to 82.6] | 82.4 [71.8 to 90.3]

7. Secondary Outcome: Magnitude of Cellular Immune Response Assessed by Number of SFC/Million PBMCs Measured by IFN-γ ELISPOT at 1 Month Post First, Pre- Second Vaccination, 1 and 6 Months Post Second Vaccination, and Annually at Years 1, 2, and 3 by Country
Description: The magnitude of cellular immune response by country was assessed by the number of SFC/million PBMCs for participants with a cellular immune response. Cellular immune response was defined as IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1) and ≥ 5 spots per well. Data (SFC/million PBMC) for participants with a cellular immune response to any peptide pool is reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2. Data is reported as per enrollment by country (Panama and Philippines).
Time Frame: as for outcome 6
Population: PPS 'by country' included all participants from the FAS who have no major protocol violations. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Median (Inter-Quartile Range); unit: SFC/million PBMCs
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Panama | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Philippines
Number analyzed (Participants) | 97 | 98
SFC/million PBMCs
  Day 30: number analyzed (Participants) | 73 | 90
  Day 30 | 1019.0 [437.0 to 2228.0] | 1065.0 [418.0 to 2546.0]
  Day 90: number analyzed (Participants) | 82 | 92
  Day 90 | 531.5 [252.0 to 1116.0] | 577.5 [255.5 to 1396.0]
  Day 120: number analyzed (Participants) | 73 | 95
  Day 120 | 780.0 [322.0 to 1525.0] | 1003.0 [437.0 to 2304.0]
  Day 270: number analyzed (Participants) | 71 | 94
  Day 270 | 426.0 [184.0 to 1382.0] | 512.5 [210.0 to 1130.0]
  Year 1: number analyzed (Participants) | 76 | 82
  Year 1 | 209.0 [81.5 to 494.0] | 178.5 [73.0 to 451.0]
  Year 2: number analyzed (Participants) | 45 | 81
  Year 2 | 76.0 [45.0 to 229.0] | 124.0 [41.0 to 615.0]
  Year 3: number analyzed (Participants) | 63 | 70
  Year 3 | 147.0 [51.0 to 280.0] | 117.0 [43.0 to 659.0]

8. Secondary Outcome: Magnitude of Cellular Immune Response Assessed by Number of SFC/Million PBMCs Measured by IFN-γ ELISPOT 1Month Post First Vaccination,Pre-second Vaccination;1,6Months Post Second Vaccination, Annually at Years1,2,3 by Dengue Baseline Seropositivity Status
Description: The magnitude of cellular immune response by dengue Baseline seropositivity status was assessed by the number of SFC/million PBMCs for participants with a cellular immune response. Cellular immune response was defined as IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1) and ≥ 5 spots per well. Seropositive at Baseline was defined as a reciprocal neutralizing titer >=10 for one or more dengue serotypes. Seronegative at Baseline was defined as having a reciprocal neutralizing titer <10 for all dengue serotypes. The 4 dengue virus serotypes were dengue virus (DENV)-1, DENV-2, DENV-3 and DENV-4. Cellular immune response to any peptide pool was reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2. Data is reported per Baseline seropositivity status of participants (Seropositive and Seronegative).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SFC/million PBMCs
Groups:
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: Seronegative: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants seronegative at Baseline.
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Seropositive | Tetravalent Dengue Vaccine (TDV) 0.5 mL: Seronegative
Number analyzed (Participants) | 109 | 86
SFC/million PBMCs
  Day 30: number analyzed (Participants) | 89 | 74
  Day 30 | 1415.0 [529.0 to 3302.0] | 840.5 [379.0 to 1844.0]
  Day 90: number analyzed (Participants) | 97 | 77
  Day 90 | 743.0 [257.0 to 1560.0] | 473.0 [246.0 to 927.0]
  Day 120: number analyzed (Participants) | 96 | 72
  Day 120 | 1086.0 [429.0 to 2521.0] | 700.0 [343.0 to 1476.0]
  Day 270: number analyzed (Participants) | 94 | 71
  Day 270 | 592.5 [184.0 to 1569.0] | 400.0 [225.0 to 808.0]
  Year 1: number analyzed (Participants) | 86 | 72
  Year 1 | 275.0 [105.0 to 690.0] | 132.0 [69.0 to 247.0]
  Year 2: number analyzed (Participants) | 75 | 51
  Year 2 | 135.0 [46.0 to 615.0] | 74.0 [38.0 to 304.0]
  Year 3: number analyzed (Participants) | 72 | 61
  Year 3 | 180.0 [61.0 to 645.5] | 103.0 [35.0 to 430.0]

9. Secondary Outcome: Percentage of Participants With Cellular Immune Response to TDV in Participants >10 Years of Age
Description: Percentage of participants with cellular immune response in participants >10 years of age were reported. Cellular immune response was defined as an IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1 [M0]) and >=5 spots per well. Cellular immune response to any peptide pool was reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2.
Time Frame: Day 14
Population: PPS with participants >10 years of age included all participants from the FAS who have no major protocol violations and are >10 years of age. The overall number of participants analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 10
percentage of participants | 70.0 [34.8 to 93.3]

10. Secondary Outcome: Magnitude of Cellular Immune Response Assessed by Number of SFC/Million PBMCs Measured by IFN-γ ELISPOT in Participants >10 Years of Age
Description: The magnitude of cellular immune response was assessed by the number of SFC/million PBMCs for participants with a cellular immune response. Cellular immune response was defined as IFN-γ ELISPOT response that was >3 times higher compared to Baseline (Day 1) and ≥ 5 spots per well. Cellular immune response to any peptide pool was reported. The peptide pool included NS3 and NS5 for each of the dengue serotype: DENV-1, DENV-2, DENV-3 and DENV-4 and NS1 for DENV-2. SFC/million PBMC for any peptide pool is reported in participants >10 years of age.
Time Frame: Day 14
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: SFC/million PBMCs
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 7
SFC/million PBMCs | 227.0 [124.0 to 3781.0]

11. Secondary Outcome: Phenotype Characterization of Cellular Immune Response Assessed by Percentage of Total T Cells of Cellular Response to DENV-2 NS Peptides at 1Month Post First Vaccination,Pre-second Vaccination;1,6Months Post Second Vaccination, Annually at Years1,2,3
Description: The phenotype characterization of cellular immune response was assessed by intracellular cytokine staining (ICS) by the frequency of total cluster of differentiation 4 (CD4)+ and CD8+ T cells and was performed in a subset of participants with IFN- γ ELISPOT responses >500 SFC/million cells and availability of sufficient cells. The peptide pools included NS1, NS3 and NS5 for DENV-2 serotype. Data are presented for the different expression profiles of interferon-gamma (IFN-γ), interleukin-2 (IL-2) and tumor necrosis factor-alpha (TNF-α) cytokines for each peptide pool. Data is reported based on the type of T cells present in participants at the time of analysis (CD4+ T cells and CD8+ T cells).
Time Frame: as for outcome 6
Population: ICS Subset 'by T-cells' included participants from PPS who have IFN-γ ELISPOT responses >500 SFC/million PBMCs and availability of sufficient cells. Number analyzed is the number of participants with data available for analysis for specific category.
Measure: Median (Inter-Quartile Range); unit: percentage of T cells
Groups:
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: CD4+ T Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): CD4+ T cells.
- Tetravalent Dengue Vaccine (TDV) 0.5 mL: CD8+ T Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): CD8+ T cells.
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL: CD4+ T Cells | Tetravalent Dengue Vaccine (TDV) 0.5 mL: CD8+ T Cells
Number analyzed (Participants) | 79 | 79
percentage of T cells
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 30 | 0.008260 [0.003050 to 0.020000] | 0.001350 [0.000000 to 0.008190]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 30 | 0.005110 [0.001953 to 0.010000] | 0.020000 [0.002580 to 0.039350]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 30 | 0.005380 [0.002430 to 0.009420] | 0.015580 [0.003084 to 0.043000]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 30 | 0.000000 [0.000000 to 0.001350] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 30 | 0.000000 [0.000000 to 0.000130] | 0.001210 [0.000000 to 0.003000]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 30 | 0.000000 [0.000000 to 0.000120] | 0.001610 [0.000000 to 0.004370]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 30 | 0.003720 [0.000580 to 0.006770] | 0.018180 [0.000190 to 0.054000]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 30 | 0.002810 [0.000130 to 0.006420] | 0.140000 [0.058000 to 0.448100]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 30 | 0.002890 [0.000020 to 0.006240] | 0.140790 [0.028940 to 0.382000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 30 | 0.002310 [0.000000 to 0.007080] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 30 | 0.002110 [0.000000 to 0.007290] | 0.000000 [0.000000 to 0.000760]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 30 | 0.003350 [0.000000 to 0.008360] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 30 | 0.000850 [0.000000 to 0.004190] | 0.007490 [0.002150 to 0.032580]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 30 | 0.000000 [0.000000 to 0.002890] | 0.061520 [0.025260 to 0.208580]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 30 | 0.000498 [0.000000 to 0.003520] | 0.063490 [0.020000 to 0.222230]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 30 | 0.001000 [0.000000 to 0.009000] | 0.002000 [0.000000 to 0.008000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 30 | 0.000000 [0.000000 to 0.007000] | 0.000000 [0.000000 to 0.008000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 30 | 0.000000 [0.000000 to 0.010000] | 0.001700 [0.000000 to 0.010000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 30 | 0.000000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.013000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 30 | 0.010000 [0.000000 to 0.040000] | 0.012000 [0.000000 to 0.030000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 71 | 71
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 30 | 0.010000 [0.000000 to 0.050000] | 0.008000 [0.000000 to 0.030000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 90 | 0.003825 [0.001215 to 0.009130] | 0.000000 [0.000000 to 0.004075]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 90 | 0.002908 [0.000285 to 0.006325] | 0.005565 [0.001470 to 0.012500]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 90 | 0.002050 [0.000000 to 0.005690] | 0.004020 [0.000622 to 0.013000]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 90 | 0.000615 [0.000000 to 0.001460] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.002200] | 0.000000 [0.000000 to 0.001566]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.000980] | 0.000000 [0.000000 to 0.001865]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 90 | 0.001045 [0.000000 to 0.002805] | 0.005155 [0.000020 to 0.021160]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 90 | 0.001608 [0.000000 to 0.003055] | 0.106350 [0.032245 to 0.198546]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 90 | 0.000750 [0.000000 to 0.002583] | 0.076145 [0.017500 to 0.156850]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 90 | 0.001050 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.000884]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 90 | 0.000910 [0.000000 to 0.003360] | 0.000000 [0.000000 to 0.000340]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 72 | 71
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 90 | 0.002925 [0.000000 to 0.006000] | 0.000000 [0.000000 to 0.000374]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.001425] | 0.001820 [0.000000 to 0.006305]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.000973] | 0.022310 [0.007580 to 0.075184]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.001251] | 0.021455 [0.002945 to 0.045665]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.009000] | 0.001500 [0.000000 to 0.010000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.009000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 90 | 0.003000 [0.000000 to 0.010500] | 0.000000 [0.000000 to 0.010000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.009500]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.028500] | 0.012000 [0.000500 to 0.032470]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 72 | 72
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 90 | 0.009500 [0.000000 to 0.050000] | 0.008500 [0.000000 to 0.026500]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 120 | 0.008340 [0.003340 to 0.017000] | 0.001320 [0.000000 to 0.004240]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 120 | 0.003410 [0.001041 to 0.007190] | 0.010000 [0.002650 to 0.018000]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 120 | 0.002100 [0.000000 to 0.004710] | 0.007850 [0.002230 to 0.027000]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 120 | 0.001050 [0.000000 to 0.002420] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.001420] | 0.000000 [0.000000 to 0.001800]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 120 | 0.000000 [0.000000 to 0.000935] | 0.000960 [0.000000 to 0.002340]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 120 | 0.002110 [0.000000 to 0.005070] | 0.007340 [0.000000 to 0.029850]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 120 | 0.002000 [0.000000 to 0.004160] | 0.116110 [0.047000 to 0.317000]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 120 | 0.000860 [0.000000 to 0.002820] | 0.096230 [0.030050 to 0.207090]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 120 | 0.007160 [0.002000 to 0.015040] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.004710] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 120 | 0.003350 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 120 | 0.002070 [0.000000 to 0.005030] | 0.004080 [0.000000 to 0.011000]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 120 | 0.000990 [0.000000 to 0.002630] | 0.038000 [0.013270 to 0.094810]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 120 | 0.000000 [0.000000 to 0.002480] | 0.018850 [0.007000 to 0.060560]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 120 | 0.009000 [0.000000 to 0.014000] | 0.002000 [0.000000 to 0.014000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 120 | 0.001000 [0.000000 to 0.010000] | 0.001000 [0.000000 to 0.017000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 120 | 0.000000 [0.000000 to 0.013000] | 0.001000 [0.000000 to 0.015000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 120 | 0.002000 [0.000000 to 0.028000] | 0.004000 [0.000000 to 0.020000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.030000] | 0.012000 [0.000000 to 0.028000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 75 | 75
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 120 | 0.020000 [0.000000 to 0.050000] | 0.012000 [0.000000 to 0.030000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 270 | 0.006150 [0.002940 to 0.015000] | 0.000000 [0.000000 to 0.002450]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 270 | 0.002520 [0.000050 to 0.006570] | 0.004630 [0.001430 to 0.010157]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 270 | 0.002840 [0.000220 to 0.005230] | 0.004430 [0.000955 to 0.019000]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.000980] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001830]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001470]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 270 | 0.001100 [0.000000 to 0.003380] | 0.004620 [0.000000 to 0.023950]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 270 | 0.001210 [0.000000 to 0.003450] | 0.089000 [0.033000 to 0.213910]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 270 | 0.000334 [0.000000 to 0.002500] | 0.067000 [0.021000 to 0.197960]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 270 | 0.004010 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.004830] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 270 | 0.001630 [0.000000 to 0.005000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.002570] | 0.003060 [0.000000 to 0.008450]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.001720] | 0.015360 [0.002440 to 0.029940]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.002320] | 0.013000 [0.002000 to 0.029600]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 270 | 0.001000 [0.000000 to 0.008000] | 0.001000 [0.000000 to 0.007000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.001980] | 0.000000 [0.000000 to 0.005000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.007000] | 0.000000 [0.000000 to 0.006000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.014000] | 0.002000 [0.000000 to 0.018000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 270 | 0.005000 [0.000000 to 0.030000] | 0.015000 [0.000000 to 0.044000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 71 | 71
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.050000] | 0.014000 [0.000000 to 0.033000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 1 | 0.003980 [0.000000 to 0.007470] | 0.000000 [0.000000 to 0.001410]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 1 | 0.001998 [0.000000 to 0.005000] | 0.001360 [0.000000 to 0.003970]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 1 | 0.001275 [0.000000 to 0.005900] | 0.001600 [0.000000 to 0.006660]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 1 | 0.000105 [0.000000 to 0.001700] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.001240] | 0.000000 [0.000000 to 0.001120]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 1 | 0.000000 [0.000000 to 0.001370] | 0.000000 [0.000000 to 0.000828]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 1 | 0.001085 [0.000000 to 0.003000] | 0.000000 [0.000000 to 0.012000]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 1 | 0.001100 [0.000000 to 0.002718] | 0.022915 [0.004790 to 0.054750]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 1 | 0.000856 [0.000000 to 0.003000] | 0.022135 [0.002010 to 0.069860]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 1 | 0.003000 [0.000000 to 0.009125] | 0.000000 [0.000000 to 0.001130]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 1 | 0.001585 [0.000000 to 0.005470] | 0.000000 [0.000000 to 0.000968]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 1 | 0.003545 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.001370]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 1 | 0.000587 [0.000000 to 0.002580] | 0.000434 [0.000000 to 0.005200]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.002000] | 0.003075 [0.000000 to 0.010870]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 1 | 0.000000 [0.000000 to 0.001880] | 0.003400 [0.000000 to 0.016640]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 1 | 0.000000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.009000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 1 | 0.000500 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.008000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 1 | 0.003500 [0.000000 to 0.018000] | 0.000000 [0.000000 to 0.010000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 1 | 0.002500 [0.000000 to 0.060000] | 0.000000 [0.000000 to 0.007000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.070000] | 0.005210 [0.000000 to 0.022000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 70 | 70
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 1 | 0.042500 [0.000000 to 0.120000] | 0.007000 [0.000000 to 0.020250]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 2 | 0.002920 [0.000140 to 0.006890] | 0.000000 [0.000000 to 0.001050]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 2 | 0.000727 [0.000000 to 0.003915] | 0.001925 [0.000000 to 0.004043]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 2 | 0.001500 [0.000000 to 0.005815] | 0.001535 [0.000000 to 0.005245]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.001040] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.000853] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 2 | 0.000000 [0.000000 to 0.001435] | 0.000000 [0.000000 to 0.000982]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 2 | 0.000871 [0.000000 to 0.002065] | 0.001015 [0.000000 to 0.004355]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 2 | 0.000080 [0.000000 to 0.001760] | 0.014120 [0.004700 to 0.059078]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 2 | 0.000810 [0.000000 to 0.002310] | 0.013923 [0.002940 to 0.052000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 2 | 0.001000 [0.000000 to 0.005000] | 0.000100 [0.000000 to 0.001980]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.003405] | 0.003625 [0.001660 to 0.007235]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 2 | 0.002835 [0.000000 to 0.009205] | 0.002915 [0.000000 to 0.008730]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 2 | 0.000420 [0.000000 to 0.002115] | 0.000100 [0.000000 to 0.001980]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 2 | 0.000210 [0.000000 to 0.001285] | 0.003625 [0.001660 to 0.007235]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 2 | 0.000150 [0.000000 to 0.001500] | 0.002915 [0.000000 to 0.008730]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.001500] | 0.000000 [0.000000 to 0.005000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.002000] | 0.000000 [0.000000 to 0.003180]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 2 | 0.000000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.008500]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.039000] | 0.000000 [0.000000 to 0.001050]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 2 | 0.009500 [0.000000 to 0.055000] | 0.001295 [0.000000 to 0.017150]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 56 | 56
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 2 | 0.029500 [0.000000 to 0.105000] | 0.003000 [0.000000 to 0.017150]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 3 | 0.002450 [0.000000 to 0.005360] | 0.000000 [0.000000 to 0.001070]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 3 | 0.000696 [0.000000 to 0.006250] | 0.000950 [0.000000 to 0.004030]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 3 | 0.002510 [0.000000 to 0.006480] | 0.000856 [0.000000 to 0.005240]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.000999] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 3 | 0.000060 [0.000000 to 0.001390] | 0.000000 [0.000000 to 0.000647]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 3 | 0.000122 [0.000000 to 0.002741] | 0.000000 [0.000000 to 0.000905]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 3 | 0.000160 [0.000000 to 0.001990] | 0.000000 [0.000000 to 0.002670]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.001574] | 0.006290 [0.000930 to 0.022070]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 3 | 0.000090 [0.000000 to 0.001980] | 0.007770 [0.001000 to 0.040020]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 3 | 0.001670 [0.000000 to 0.005550] | 0.000000 [0.000000 to 0.000873]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 3 | 0.001000 [0.000000 to 0.003000] | 0.000000 [0.000000 to 0.000980]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 3 | 0.002000 [0.000000 to 0.007000] | 0.000000 [0.000000 to 0.001060]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 3 | 0.000048 [0.000000 to 0.001480] | 0.000000 [0.000000 to 0.002250]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.001310] | 0.002340 [0.000000 to 0.006260]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 3 | 0.000180 [0.000000 to 0.001630] | 0.002380 [0.000000 to 0.010000]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.005000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.009000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 3 | 0.002000 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.007000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.005000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.011000] | 0.003000 [0.000000 to 0.016000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 69 | 69
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 3 | 0.020000 [0.000000 to 0.060000] | 0.005000 [0.000000 to 0.017000]

12. Secondary Outcome: Phenotype Characterization of Cellular Immune Response Assessed by Percentage of Total T Cells of Cellular Response DENV-2 NS Peptides,1Month Post First Vaccination,Pre Second Vaccination;1,6Months Post Second Vaccination,Annually at Years1,2,3 by Country
Description: The phenotype characterization of cellular immune response by country was assessed by ICS by the frequency of total CD4+ and CD8+ T cells and was performed in a subset of participants with IFN- γ ELISPOT responses >500 SFC/million cells and availability of sufficient cells. The peptide pools included NS1, NS3 and NS5 for DENV-2 serotype. Data are presented for the different expression profiles of IFN-γ, IL-2 and TNF-α cytokines for each peptide pool. Data is reported per country (Panama and Philippines) based on the type of T cells present in participants at the time of analysis (CD4+ T cells and CD8+ T cells).
Time Frame: as for outcome 6
Population: ICS Subset 'by country based on T-cells' included participants from PPS who have IFN-γ ELISPOT responses >500 SFC/million PBMCs and availability of sufficient cells. Number analyzed is the number of participants with data available for analysis for specific category.
Measure: Median (Inter-Quartile Range); unit: percentage of T cells
Groups:
- TDV 0.5 mL: Panama: CD4+ T Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants from Panama, CD4+ T cells.
- TDV 0.5 mL: Philippines: CD4+ T Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants from Philippines, CD4+ T cells.
- TDV 0.5 mL: Panama: CD8+ T Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants from Panama, CD8+ T cells.
- TDV 0.5 ml: Philippines: CD8+ T Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants from Philippines, CD8+ T cells.
Arm/Group | TDV 0.5 mL: Panama: CD4+ T Cells | TDV 0.5 mL: Philippines: CD4+ T Cells | TDV 0.5 mL: Panama: CD8+ T Cells | TDV 0.5 ml: Philippines: CD8+ T Cells
Number analyzed (Participants) | 33 | 46 | 33 | 46
percentage of T cells
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 30 | 0.005670 [0.001120 to 0.017245] | 0.010590 [0.004880 to 0.020000] | 0.001655 [0.000000 to 0.023500] | 0.001350 [0.000000 to 0.004720]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 30 | 0.002700 [0.001651 to 0.006900] | 0.006810 [0.002040 to 0.011040] | 0.014500 [0.002155 to 0.036000] | 0.021000 [0.004490 to 0.040260]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 30 | 0.003892 [0.001960 to 0.007760] | 0.005450 [0.003160 to 0.012000] | 0.021000 [0.002955 to 0.039500] | 0.014000 [0.003084 to 0.049000]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 30 | 0.000000 [0.000000 to 0.001810] | 0.000000 [0.000000 to 0.000850] | 0.000000 [0.000000 to 0.000545] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 30 | 0.000000 [0.000000 to 0.000865] | 0.000000 [0.000000 to 0.000000] | 0.001170 [0.000000 to 0.002990] | 0.001210 [0.000000 to 0.003340]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 30 | 0.000000 [0.000000 to 0.001013] | 0.000000 [0.000000 to 0.000000] | 0.001825 [0.000000 to 0.004000] | 0.001490 [0.000000 to 0.004640]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 30 | 0.003935 [0.000208 to 0.006730] | 0.003720 [0.000740 to 0.008820] | 0.024675 [0.000530 to 0.144580] | 0.014000 [0.000190 to 0.030330]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 30 | 0.002880 [0.000202 to 0.004855] | 0.002710 [0.000130 to 0.006670] | 0.114125 [0.034725 to 0.402570] | 0.172000 [0.065720 to 0.588300]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 30 | 0.003100 [0.000195 to 0.006109] | 0.002890 [0.000010 to 0.006340] | 0.129260 [0.037645 to 0.344770] | 0.142870 [0.026180 to 0.390000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 30 | 0.001820 [0.000000 to 0.004055] | 0.004222 [0.000000 to 0.009470] | 0.000000 [0.000000 to 0.000090] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 30 | 0.002110 [0.000000 to 0.009815] | 0.001700 [0.000000 to 0.006610] | 0.000000 [0.000000 to 0.001004] | 0.000000 [0.000000 to 0.000180]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 30 | 0.003000 [0.000000 to 0.009500] | 0.003350 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 30 | 0.001440 [0.000000 to 0.004830] | 0.000850 [0.000000 to 0.003260] | 0.019265 [0.004200 to 0.078745] | 0.006850 [0.000850 to 0.015340]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 30 | 0.001240 [0.000000 to 0.002885] | 0.000000 [0.000000 to 0.003160] | 0.065510 [0.025630 to 0.162840] | 0.061520 [0.024540 to 0.287780]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 30 | 0.000620 [0.000000 to 0.003105] | 0.000498 [0.000000 to 0.003550] | 0.074245 [0.021500 to 0.190910] | 0.053520 [0.014000 to 0.230980]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 30 | 0.005000 [0.000000 to 0.012145] | 0.000000 [0.000000 to 0.004000] | 0.002000 [0.000000 to 0.010500] | 0.001620 [0.000000 to 0.008000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 30 | 0.000500 [0.000000 to 0.011645] | 0.000000 [0.000000 to 0.002000] | 0.000000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.005000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 30 | 0.008590 [0.000000 to 0.017500] | 0.000000 [0.000000 to 0.004000] | 0.007000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.008000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 30 | 0.000000 [0.000000 to 0.006000] | 0.000000 [0.000000 to 0.030000] | 0.004000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.010000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 30 | 0.004500 [0.000000 to 0.025500] | 0.010000 [0.000000 to 0.048000] | 0.008500 [0.003000 to 0.019000] | 0.014000 [0.000000 to 0.040000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 28 | 43 | 28 | 43
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 30 | 0.000000 [0.000000 to 0.040000] | 0.020000 [0.000000 to 0.050000] | 0.009000 [0.000000 to 0.024500] | 0.002000 [0.000000 to 0.035000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 90 | 0.001485 [0.000000 to 0.006030] | 0.005670 [0.002370 to 0.010370] | 0.000000 [0.000000 to 0.002070] | 0.001030 [0.000000 to 0.004850]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 90 | 0.002448 [0.000000 to 0.007030] | 0.003491 [0.000710 to 0.006290] | 0.003364 [0.000000 to 0.006120] | 0.008860 [0.003110 to 0.016000]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 90 | 0.001415 [0.000000 to 0.005600] | 0.003270 [0.000791 to 0.005780] | 0.003560 [0.001220 to 0.008740] | 0.005580 [0.000570 to 0.017770]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 90 | 0.000100 [0.000000 to 0.002130] | 0.000679 [0.000000 to 0.001300] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000722]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.002690] | 0.000515 [0.000000 to 0.001790] | 0.000000 [0.000000 to 0.001320] | 0.000837 [0.000000 to 0.001920]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.001360] | 0.000000 [0.000000 to 0.000921] | 0.000000 [0.000000 to 0.001680] | 0.001175 [0.000000 to 0.003450]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 90 | 0.000545 [0.000000 to 0.002740] | 0.001290 [0.000000 to 0.002870] | 0.003760 [0.000000 to 0.042000] | 0.005470 [0.000662 to 0.019000]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 90 | 0.000645 [0.000000 to 0.002690] | 0.002120 [0.000000 to 0.003770] | 0.047980 [0.027290 to 0.154680] | 0.125320 [0.058820 to 0.213810]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.001810] | 0.001120 [0.000000 to 0.003650] | 0.077000 [0.015630 to 0.158700] | 0.067000 [0.021020 to 0.155000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.001010] | 0.004140 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000950]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 90 | 0.000793 [0.000000 to 0.003000] | 0.001000 [0.000000 to 0.004230] | 0.000000 [0.00000 to 0.00000] | 0.00000 [0.00000 to 0.000791]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 90 | 0.001000 [0.000000 to 0.003000] | 0.004530 [0.001220 to 0.008000] | 0.00000 [0.00000 to 0.00000] | 0.00000 [0.00000 to 0.000725]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.002120] | 0.000000 [0.000000 to 0.000968] | 0.003210 [0.000000 to 0.019000] | 0.001540 [0.000000 to 0.004780]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.001680] | 0.000000 [0.000000 to 0.000742] | 0.018000 [0.001000 to 0.063760] | 0.037000 [0.011370 to 0.080257]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.002290] | 0.000000 [0.000000 to 0.000949] | 0.020970 [0.003000 to 0.059000] | 0.021940 [0.002890 to 0.036310]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.008000] | 0.002000 [0.000000 to 0.011000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 90 | 0.004000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.007000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 90 | 0.007000 [0.000000 to 0.011000] | 0.002000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.015000] | 0.000000 [0.000000 to 0.010000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.050000] | 0.000000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.009000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.019000] | 0.000000 [0.000000 to 0.036000] | 0.004000 [0.000000 to 0.022000] | 0.020000 [0.002000 to 0.042000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 31 | 41 | 31 | 41
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.030000] | 0.026000 [0.000000 to 0.060000] | 0.005000 [0.000000 to 0.017000] | 0.010000 [0.000000 to 0.030000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 120 | 0.005531 [0.003340 to 0.012780] | 0.009230 [0.003860 to 0.018610] | 0.001590 [0.000000 to 0.006910] | 0.001100 [0.000000 to 0.002580]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 120 | 0.002690 [0.001041 to 0.007190] | 0.003495 [0.001420 to 0.006660] | 0.010000 [0.002850 to 0.016000] | 0.010000 [0.002650 to 0.019000]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 120 | 0.000661 [0.000000 to 0.002990] | 0.002598 [0.000000 to 0.005470] | 0.013000 [0.004830 to 0.021000] | 0.006905 [0.001180 to 0.028000]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 120 | 0.000900 [0.000000 to 0.002580] | 0.001135 [0.000000 to 0.002180] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001670] | 0.000000 [0.000000 to 0.001440] | 0.000000 [0.000000 to 0.001920]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 120 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001190] | 0.000000 [0.000000 to 0.001650] | 0.001175 [0.000000 to 0.003450]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 120 | 0.002396 [0.000260 to 0.005000] | 0.002045 [0.000000 to 0.005070] | 0.011000 [0.001100 to 0.066340] | 0.005500 [0.000000 to 0.019000]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 120 | 0.002456 [0.000250 to 0.005980] | 0.001800 [0.000000 to 0.003200] | 0.092920 [0.038250 to 0.160000] | 0.153500 [0.048520 to 0.353170]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 120 | 0.001590 [0.000000 to 0.002636] | 0.000702 [0.000000 to 0.002960] | 0.094740 [0.030050 to 0.205000] | 0.096615 [0.031580 to 0.220000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 120 | 0.005710 [0.000000 to 0.010000] | 0.008335 [0.002900 to 0.017000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.005520] | 0.000000 [0.000000 to 0.004000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 120 | 0.003580 [0.000000 to 0.008000] | 0.003275 [0.000000 to 0.010660] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001250]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 120 | 0.002490 [0.000000 to 0.005560] | 0.001520 [0.000000 to 0.004380] | 0.006000 [0.001770 to 0.019000] | 0.003750 [0.000000 to 0.007240]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 120 | 0.001620 [0.000000 to 0.002630] | 0.000365 [0.000000 to 0.002000] | 0.033420 [0.009000 to 0.081860] | 0.039000 [0.015000 to 0.104850]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 120 | 0.000000 [0.000000 to 0.002000] | 0.000205 [0.000000 to 0.002830] | 0.022820 [0.012340 to 0.058000] | 0.018425 [0.004130 to 0.060560]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 120 | 0.010000 [0.000000 to 0.015000] | 0.007000 [0.000000 to 0.012000] | 0.000000 [0.000000 to 0.008000] | 0.002000 [0.000000 to 0.017000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.005000] | 0.001500 [0.000000 to 0.011000] | 0.005000 [0.000000 to 0.017000] | 0.000000 [0.000000 to 0.012000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 120 | 0.001000 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.013000] | 0.005000 [0.000000 to 0.015000] | 0.000000 [0.000000 to 0.014000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 120 | 0.001000 [0.000000 to 0.020000] | 0.002000 [0.000000 to 0.030000] | 0.004000 [0.000000 to 0.017000] | 0.003000 [0.000000 to 0.020000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.030000] | 0.000000 [0.000000 to 0.028000] | 0.010000 [0.000000 to 0.020000] | 0.016500 [0.000000 to 0.033000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 29 | 46 | 29 | 46
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 120 | 0.020000 [0.000000 to 0.050000] | 0.015000 [0.000000 to 0.049000] | 0.013000 [0.000000 to 0.027340] | 0.011000 [0.000000 to 0.031000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 270 | 0.006400 [0.002940 to 0.015180] | 0.005090 [0.002935 to 0.014500] | 0.000000 [0.000000 to 0.003850] | 0.000000 [0.000000 to 0.002285]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 270 | 0.004470 [0.001750 to 0.007780] | 0.001540 [0.000000 to 0.004138] | 0.002920 [0.000020 to 0.014000] | 0.005090 [0.001570 to 0.009779]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 270 | 0.002890 [0.001910 to 0.004530] | 0.002393 [0.000000 to 0.005765] | 0.006040 [0.001120 to 0.030780] | 0.003620 [0.000478 to 0.014160]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.001490] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.002100] | 0.000000 [0.000000 to 0.000915]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.001220] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001220] | 0.000000 [0.000000 to 0.001550]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 270 | 0.000200 [0.000000 to 0.002270] | 0.001386 [0.000000 to 0.003795] | 0.004620 [0.001270 to 0.041450] | 0.004695 [0.000000 to 0.019500]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 270 | 0.002270 [0.000000 to 0.005380] | 0.000740 [0.000000 to 0.002175] | 0.073630 [0.033000 to 0.140000] | 0.099370 [0.034095 to 0.273535]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.001870] | 0.000430 [0.000000 to 0.002875] | 0.093000 [0.022090 to 0.197960] | 0.056525 [0.017440 to 0.183385]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 270 | 0.002000 [0.000000 to 0.012000] | 0.005400 [0.001685 to 0.009780] | 0.000000 [0.000000 to 0.000660] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.005400] | 0.000660 [0.000000 to 0.004630] | 0.000000 [0.000000 to 0.001160] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.004000] | 0.001955 [0.000000 to 0.006600] | 0.000000 [0.000000 to 0.001350] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.002780] | 0.000000 [0.000000 to 0.002015] | 0.004600 [0.000000 to 0.011000] | 0.001669 [0.000000 to 0.007810]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 32 | 44 | 27 | 44
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.002760] | 0.000002 [0.000000 to 0.001615] | 0.015000 [0.004570 to 0.028280] | 0.016169 [0.001670 to 0.047810]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 32 | 44 | 27 | 44
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.003550] | 0.000000 [0.000000 to 0.001285] | 0.018200 [0.006240 to 0.035000] | 0.009090 [0.000030 to 0.025060]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.008000] | 0.001000 [0.000000 to 0.007620] | 0.002000 [0.000000 to 0.009000] | 0.000500 [0.000000 to 0.005680]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.003000] | 0.001000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.001500]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.007000] | 0.000000 [0.000000 to 0.007950] | 0.000000 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.006000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.020000] | 0.005000 [0.000000 to 0.021000] | 0.000000 [0.000000 to 0.015000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.029000] | 0.005500 [0.000000 to 0.038500] | 0.016000 [0.000000 to 0.040000] | 0.010000 [0.000000 to 0.053000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 27 | 44 | 27 | 44
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.050000] | 0.000000 [0.000000 to 0.040000] | 0.021000 [0.000000 to 0.045000] | 0.010000 [0.000000 to 0.029000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 1 | 0.002825 [0.000000 to 0.008700] | 0.004303 [0.000000 to 0.007260] | 0.000000 [0.000000 to 0.001720] | 0.000000 [0.000000 to 0.001160]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 1 | 0.001835 [0.000000 to 0.006990] | 0.002138 [0.000000 to 0.004780] | 0.001970 [0.000005 to 0.004610] | 0.000000 [0.000000 to 0.003536]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 1 | 0.001486 [0.000000 to 0.004375] | 0.000538 [0.000000 to 0.006780] | 0.004090 [0.000000 to 0.010820] | 0.000935 [0.000000 to 0.004230]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 1 | 0.000758 [0.000000 to 0.002335] | 0.000000 [0.000000 to 0.001590] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 1 | 0.000035 [0.000000 to 0.001690] | 0.000000 [0.000000 to 0.001140] | 0.000000 [0.000000 to 0.000918] | 0.000000 [0.000000 to 0.001140]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 1 | 0.000000 [0.000000 to 0.001230] | 0.000000 [0.000000 to 0.001620] | 0.000000 [0.000000 to 0.000950] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 1 | 0.000004 [0.000000 to 0.002130] | 0.001599 [0.000010 to 0.005810] | 0.001650 [0.000000 to 0.025930] | 0.000000 [0.000000 to 0.001790]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 1 | 0.001170 [0.000000 to 0.002050] | 0.000965 [0.000000 to 0.003340] | 0.022915 [0.008465 to 0.046500] | 0.022820 [0.004000 to 0.061950]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 1 | 0.001065 [0.000000 to 0.001825] | 0.000766 [0.000000 to 0.003750] | 0.045815 [0.009695 to 0.094410] | 0.009520 [0.000000 to 0.036130]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 1 | 0.002758 [0.000000 to 0.007000] | 0.003735 [0.000000 to 0.011820] | 0.000000 [0.000000 to 0.001010] | 0.000000 [0.000000 to 0.001590]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.003000] | 0.003000 [0.000000 to 0.008620] | 0.000000 [0.000000 to 0.000035] | 0.000000 [0.000000 to 0.001370]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 1 | 0.001053 [0.000000 to 0.006000] | 0.004910 [0.000060 to 0.014000] | 0.000000 [0.000000 to 0.001315] | 0.000795 [0.000000 to 0.001510]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 1 | 0.000477 [0.000000 to 0.002413] | 0.000788 [0.000000 to 0.002670] | 0.002995 [0.000000 to 0.009535] | 0.000000 [0.000000 to 0.003210]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.001311] | 0.000000 [0.000000 to 0.002250] | 0.004390 [0.001090 to 0.012525] | 0.002250 [0.000000 to 0.008910]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 1 | 0.000456 [0.000000 to 0.002790] | 0.000000 [0.000000 to 0.001440] | 0.008865 [0.002510 to 0.019285] | 0.000465 [0.000000 to 0.006390]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 1 | 0.000000 [0.000000 to 0.011000] | 0.002000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.009440] | 0.000500 [0.000000 to 0.009000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.010000] | 0.001000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.004175] | 0.000000 [0.000000 to 0.008000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 1 | 0.000000 [0.000000 to 0.014500] | 0.005000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.013940] | 0.000500 [0.000000 to 0.009000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 1 | 0.000000 [0.000000 to 0.021000] | 0.020000 [0.000000 to 0.130000] | 0.000000 [0.000000 to 0.003000] | 0.000895 [0.000000 to 0.009000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.023500] | 0.025500 [0.000000 to 0.100000] | 0.003500 [0.000000 to 0.012500] | 0.010500 [0.000000 to 0.026000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 32 | 38 | 32 | 38
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 1 | 0.006500 [0.000000 to 0.085000] | 0.075000 [0.000000 to 0.180000] | 0.005500 [0.000000 to 0.018210] | 0.010000 [0.000000 to 0.022000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 2 | 0.003832 [0.001292 to 0.007035] | 0.002406 [0.000000 to 0.006890] | 0.000000 [0.000000 to 0.001050] | 0.000000 [0.000000 to 0.000998]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 2 | 0.001452 [0.000337 to 0.005767] | 0.000503 [0.000000 to 0.002644] | 0.002230 [0.000484 to 0.002745] | 0.001875 [0.000000 to 0.004790]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 2 | 0.002005 [0.000323 to 0.007710] | 0.001335 [0.000000 to 0.005545] | 0.002595 [0.001290 to 0.005245] | 0.000812 [0.000000 to 0.005740]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 2 | 0.001005 [0.000000 to 0.002250] | 0.000000 [0.000000 to 0.000797] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 2 | 0.000982 [0.000000 to 0.002760] | 0.000000 [0.000000 to 0.000007] | 0.000000 [0.000000 to 0.001062] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 2 | 0.000631 [0.000000 to 0.005337] | 0.000000 [0.000000 to 0.000743] | 0.000000 [0.000000 to 0.000988] | 0.000000 [0.000000 to 0.000982]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 2 | 0.000261 [0.000000 to 0.001360] | 0.001095 [0.000000 to 0.002335] | 0.002010 [0.000025 to 0.004425] | 0.000000 [0.000000 to 0.004290]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 2 | 0.000413 [0.000000 to 0.001012] | 0.000050 [0.000000 to 0.002470] | 0.012063 [0.003120 to 0.045755] | 0.015970 [0.006810 to 0.069945]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 2 | 0.000656 [0.000000 to 0.001710] | 0.001055 [0.000000 to 0.003220] | 0.018930 [0.008160 to 0.050495] | 0.009770 [0.002160 to 0.054000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 2 | 0.000895 [0.000000 to 0.003615] | 0.001000 [0.000000 to 0.005000] | 0.000000 [0.000000 to 0.000535] | 0.000000 [0.000000 to 0.000054]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.002060] | 0.000380 [0.000000 to 0.003775] | 0.000000 [0.000000 to 0.000927] | 0.000000 [0.000000 to 0.000908]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 2 | 0.001555 [0.000000 to 0.008615] | 0.003865 [0.000000 to 0.009705] | 0.000000 [0.000000 to 0.000856] | 0.000000 [0.000000 to 0.000963]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 2 | 0.000702 [0.000000 to 0.002704] | 0.000020 [0.000000 to 0.001690] | 0.000860 [0.000000 to 0.001435] | 0.000030 [0.000000 to 0.002080]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 2 | 0.001005 [0.000000 to 0.001785] | 0.000050 [0.000000 to 0.001196] | 0.004335 [0.002185 to 0.008140] | 0.003555 [0.000850 to 0.007200]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 2 | 0.000985 [0.000000 to 0.001820] | 0.000085 [0.000000 to 0.001405] | 0.005735 [0.002780 to 0.016800] | 0.001155 [0.000000 to 0.007580]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.000500] | 0.000000 [0.000000 to 0.003500] | 0.000000 [0.000000 to 0.006325] | 0.000000 [0.000000 to 0.005000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.003500] | 0.000000 [0.000000 to 0.002000] | 0.002180 [0.000000 to 0.006000] | 0.000000 [0.000000 to 0.001500]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 2 | 0.000500 [0.000000 to 0.022000] | 0.000000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.004385] | 0.000000 [0.000000 to 0.009500]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.020000] | 0.003500 [0.000000 to 0.044500] | 0.000000 [0.000000 to 0.002870] | 0.000000 [0.000000 to 0.001000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.030500] | 0.020000 [0.000000 to 0.070000] | 0.004155 [0.000000 to 0.013150] | 0.001295 [0.000000 to 0.019500]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 16 | 40 | 16 | 40
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 2 | 0.000500 [0.000000 to 0.065000] | 0.047000 [0.005500 to 0.110000] | 0.001370 [0.000000 to 0.013650] | 0.003500 [0.000000 to 0.020000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 3 | 0.001810 [0.000000 to 0.007589] | 0.002624 [0.000000 to 0.005010] | 0.000000 [0.000000 to 0.001030] | 0.000000 [0.000000 to 0.001240]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 3 | 0.000530 [0.000000 to 0.003668] | 0.000760 [0.000000 to 0.007520] | 0.000985 [0.000000 to 0.004030] | 0.000844 [0.000000 to 0.006500]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 3 | 0.001915 [0.000000 to 0.006970] | 0.002884 [0.000000 to 0.006480] | 0.001735 [0.000000 to 0.006330] | 0.000000 [0.000000 to 0.002690]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.000819] | 0.000000 [0.000000 to 0.001137] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.001238] | 0.000080 [0.000000 to 0.001660] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000763]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 3 | 0.001265 [0.000000 to 0.003710] | 0.000000 [0.000000 to 0.001990] | 0.000000 [0.000000 to 0.001150] | 0.000000 [0.000000 to 0.000905]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 3 | 0.000070 [0.000000 to 0.001840] | 0.000540 [0.000000 to 0.002410] | 0.001065 [0.000000 to 0.006760] | 0.000000 [0.000000 to 0.002140]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.001140] | 0.000000 [0.000000 to 0.001800] | 0.007670 [0.002000 to 0.016000] | 0.005610 [0.000600 to 0.025430]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 3 | 0.000000 [0.000000 to 0.001120] | 0.001050 [0.000000 to 0.002940] | 0.011465 [0.000000 to 0.045060] | 0.005570 [0.001000 to 0.028163]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 3 | 0.001695 [0.000000 to 0.004320] | 0.001650 [0.000000 to 0.005570] | 0.000000 [0.000000 to 0.001013] | 0.000000 [0.000000 to 0.000873]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 3 | 0.001000 [0.000000 to 0.003000] | 0.001000 [0.000000 to 0.002680] | 0.000000 [0.000000 to 0.001090] | 0.000000 [0.000000 to 0.000813]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 3 | 0.002695 [0.000000 to 0.006000] | 0.001330 [0.000000 to 0.009330] | 0.000000 [0.000000 to 0.001470] | 0.000000 [0.000000 to 0.000617]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.001219] | 0.000300 [0.000000 to 0.001630] | 0.001048 [0.000000 to 0.002680] | 0.000000 [0.000000 to 0.001950]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 3 | 0.000025 [0.000000 to 0.001630] | 0.000000 [0.000000 to 0.001310] | 0.001680 [0.000000 to 0.007000] | 0.002390 [0.000000 to 0.006260]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 3 | 0.000012 [0.000000 to 0.001820] | 0.000584 [0.000000 to 0.001560] | 0.002050 [0.000000 to 0.013360] | 0.002380 [0.000857 to 0.010000]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.006000] | 0.000000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.005000] | 0.000000 [0.000000 to 0.005000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.005000] | 0.001000 [0.000000 to 0.011000] | 0.001000 [0.000000 to 0.019000] | 0.000000 [0.000000 to 0.007000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 3 | 0.002000 [0.000000 to 0.020000] | 0.002000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.006000] | 0.001000 [0.000000 to 0.007000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.016000] | 0.000500 [0.000000 to 0.011710] | 0.000000 [0.000000 to 0.003000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.010000] | 0.001000 [0.000000 to 0.009000] | 0.008000 [0.000000 to 0.022000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 30 | 39 | 30 | 39
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 3 | 0.021500 [0.000000 to 0.050000] | 0.020000 [0.000000 to 0.090000] | 0.008500 [0.000000 to 0.017000] | 0.004000 [0.000000 to 0.015000]

13. Secondary Outcome: Phenotype Characterization of Cellular Immune Response by Percentage of Total T Cells DENV-2 NS Peptides at 1Month Post First Vaccination,Pre Second Vaccination;1,6Months Post Second Vaccination,Annually at Years1,2,3 by Dengue Baseline Seropositivity
Description: The phenotype characterization of cellular immune response by dengue Baseline seropositivity status was assessed by the frequency of total CD4+ and CD8+ T cells and was performed in a subset of participants with IFN- γ ELISPOT responses >500 SFC/million cells and availability of sufficient cells. Seropositive was defined as a reciprocal neutralizing titer (MNT50) >=10 for one or more dengue serotypes. Seronegative was defined as titer value of <10 for all 4 serotypes. The peptide pools included NS1, NS3 and NS5 for DENV-2 serotype. Data are presented for the different expression profiles of IFN-γ, IL-2 and TNF-α cytokines for each peptide pool. Data is reported per Baseline seropositivity status (Seropositive and Seronegative) based on the type of T cells present in participants at the time of analysis (CD4+ T cells and CD8+ T cells).
Time Frame: as for outcome 6
Population: ICS Subset 'by Baseline seropositivity status based on T-cells' included participants from PPS who have IFN-γ ELISPOT responses >500 SFC/million PBMCs and availability of sufficient cells. Number analyzed=participants with data available for analysis for specific category.
Measure: Median (Inter-Quartile Range); unit: percentage of T cells
Groups:
- TDV 0.5 mL: Seropositive: CD4+ T-Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants seropositive at Baseline, CD4+ T cells.
- TDV 0.5 mL: Seronegative: CD4+ T-Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants seronegative at Baseline, CD4+ T cells.
- TDV 0.5 mL: Seropositive: CD8+ T- Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants seropositive at Baseline, CD8+ T cells.
- TDV 0.5 mL: Seronegative: CD8+ T-Cells: TDV 0.5 mL, SC injection, on Day 1 (Month 0) and Day 90 (Month 3): Participants seronegative at Baseline, CD8+ T cells.
Arm/Group | TDV 0.5 mL: Seropositive: CD4+ T-Cells | TDV 0.5 mL: Seronegative: CD4+ T-Cells | TDV 0.5 mL: Seropositive: CD8+ T- Cells | TDV 0.5 mL: Seronegative: CD8+ T-Cells
Number analyzed (Participants) | 44 | 35 | 44 | 35
percentage of T cells
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 30 | 0.013000 [0.004820 to 0.023000] | 0.007655 [0.001679 to 0.011295] | 0.002170 [0.000000 to 0.007600] | 0.000245 [0.000000 to 0.009595]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 30 | 0.005140 [0.001960 to 0.014000] | 0.004985 [0.001651 to 0.008985] | 0.021000 [0.002540 to 0.039350] | 0.017000 [0.003855 to 0.038500]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 30 | 0.005380 [0.002410 to 0.012000] | 0.005255 [0.002660 to 0.009030] | 0.018000 [0.002380 to 0.050000] | 0.009560 [0.003965 to 0.028500]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 30 | 0.000000 [0.000000 to 0.001300] | 0.000000 [0.000000 to 0.001475] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 30 | 0.000000 [0.000000 to 0.001060] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.003340] | 0.001330 [0.000000 to 0.002990]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 30 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001100] | 0.001540 [0.000000 to 0.004160] | 0.001695 [0.000000 to 0.004990]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 30 | 0.004740 [0.000930 to 0.008483] | 0.003070 [0.000398 to 0.005920] | 0.018190 [0.000000 to 0.066470] | 0.015540 [0.001500 to 0.051595]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 30 | 0.002710 [0.000000 to 0.006750] | 0.002885 [0.000779 to 0.005040] | 0.108250 [0.052230 to 0.490000] | 0.168175 [0.063270 to 0.431355]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 30 | 0.002630 [0.001070 to 0.005530] | 0.003785 [0.000000 to 0.007035] | 0.150000 [0.034000 to 0.307000] | 0.117545 [0.027560 to 0.490450]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 30 | 0.003620 [0.000000 to 0.011000] | 0.002275 [0.000000 to 0.006070] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000008]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 30 | 0.002150 [0.000000 to 0.008000] | 0.001230 [0.000000 to 0.004635] | 0.000000 [0.000000 to 0.000310] | 0.000000 [0.000000 to 0.001035]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 30 | 0.003720 [0.000000 to 0.007610] | 0.002270 [0.000000 to 0.009435] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000488]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 30 | 0.000850 [0.000000 to 0.003640] | 0.000835 [0.000000 to 0.004635] | 0.007750 [0.002150 to 0.035143] | 0.007370 [0.002315 to 0.030290]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 30 | 0.000000 [0.000000 to 0.003160] | 0.000065 [0.000000 to 0.002450] | 0.065380 [0.013470 to 0.170000] | 0.051500 [0.029850 to 0.238910]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 30 | 0.000280 [0.000000 to 0.002940] | 0.000900 [0.000000 to 0.004040] | 0.053520 [0.022000 to 0.116020] | 0.101275 [0.017460 to 0.234760]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 30 | 0.001000 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.009590] | 0.002000 [0.000000 to 0.008000] | 0.002000 [0.000000 to 0.009500]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 30 | 0.000000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.003500] | 0.000000 [0.000000 to 0.007730] | 0.000000 [0.000000 to 0.008110]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 30 | 0.000000 [0.000000 to 0.010000] | 0.000500 [0.000000 to 0.009090] | 0.000000 [0.000000 to 0.010000] | 0.003610 [0.000000 to 0.009500]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 30 | 0.003000 [0.000000 to 0.030000] | 0.000000 [0.000000 to 0.007000] | 0.005000 [0.000000 to 0.018000] | 0.000000 [0.000000 to 0.004500]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 30 | 0.010000 [0.000000 to 0.045000] | 0.001500 [0.000000 to 0.030000] | 0.018000 [0.003000 to 0.035000] | 0.006000 [0.000000 to 0.020000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 30: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 30 | 0.028000 [0.000000 to 0.070000] | 0.000000 [0.000000 to 0.031000] | 0.015000 [0.000000 to 0.032000] | 0.000000 [0.000000 to 0.024500]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 90 | 0.005720 [0.002968 to 0.010690] | 0.002190 [0.001020 to 0.006030] | 0.000013 [0.000000 to 0.004300] | 0.000000 [0.000000 to 0.002980]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 90 | 0.003592 [0.000811 to 0.007360] | 0.001325 [0.000000 to 0.005820] | 0.004660 [0.001440 to 0.013770] | 0.005880 [0.001600 to 0.008860]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 90 | 0.002795 [0.000000 to 0.006900] | 0.001420 [0.000000 to 0.005530] | 0.003260 [0.000000 to 0.014000] | 0.004563 [0.001490 to 0.009010]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 90 | 0.000842 [0.000000 to 0.001960] | 0.000000 [0.000000 to 0.000888] | 0.000000 [0.000000 to 0.000722] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 90 | 0.000544 [0.000000 to 0.002510] | 0.000000 [0.000000 to 0.000824] | 0.000785 [0.000000 to 0.002560] | 0.000000 [0.000000 to 0.001132]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.000921] | 0.000000 [0.000000 to 0.001039] | 0.000383 [0.000000 to 0.001620] | 0.000000 [0.000000 to 0.002050]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 90 | 0.001540 [0.000000 to 0.003473] | 0.000490 [0.000000 to 0.001370] | 0.002893 [0.000040 to 0.019000] | 0.006540 [0.000000 to 0.024660]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 90 | 0.001583 [0.000000 to 0.003050] | 0.001810 [0.000000 to 0.003060] | 0.103350 [0.034000 to 0.213810] | 0.107000 [0.031000 to 0.178620]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 90 | 0.001090 [0.000000 to 0.003265] | 0.000410 [0.000000 to 0.002460] | 0.081000 [0.012110 to 0.129362] | 0.069105 [0.019340 to 0.192000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 90 | 0.001245 [0.000000 to 0.007850] | 0.001050 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.000912] | 0.000000 [0.000000 to 0.000650]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.002770] | 0.001880 [0.000000 to 0.004000] | 0.000000 [0.000000 to 0.000791] | 0.000000 [0.000000 to 0.000030]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 90 | 0.003980 [0.000000 to 0.006330] | 0.002055 [0.000000 to 0.005370] | 0.000000 [0.000000 to 0.000022] | 0.000000 [0.000000 to 0.000725]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 90 | 0.000010 [0.000000 to 0.001830] | 0.000000 [0.000000 to 0.001080] | 0.002390 [0.000000 to 0.006940] | 0.001535 [0.000000 to 0.005310]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.001070] | 0.000000 [0.000000 to 0.000860] | 0.039000 [0.009950 to 0.096152] | 0.017000 [0.006240 to 0.043000]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.001520] | 0.000000 [0.000000 to 0.000949] | 0.026425 [0.002250 to 0.059000] | 0.015420 [0.004490 to 0.041610]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.009000] | 0.000500 [0.000000 to 0.008000] | 0.002000 [0.000000 to 0.006000] | 0.000500 [0.000000 to 0.012000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.009000] | 0.002000 [0.000000 to 0.010000] | 0.000500 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.011000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 90 | 0.001500 [0.000000 to 0.010000] | 0.006500 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.009000] | 0.001000 [0.000000 to 0.011000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 90 | 0.000000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.008000] | 0.000000 [0.000000 to 0.012000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 90 | 0.000000 [0.000000 to 0.036000] | 0.001000 [0.000000 to 0.020000] | 0.008405 [0.001000 to 0.038000] | 0.018000 [0.000000 to 0.032000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 90: number analyzed (Participants) | 38 | 34 | 38 | 34
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 90 | 0.000000 [0.000000 to 0.050000] | 0.010405 [0.000000 to 0.050000] | 0.005450 [0.000000 to 0.027000] | 0.009500 [0.000000 to 0.026000]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 120 | 0.011000 [0.003860 to 0.017000] | 0.005531 [0.003340 to 0.016010] | 0.001400 [0.000000 to 0.004030] | 0.001320 [0.000000 to 0.004240]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 120 | 0.003480 [0.000000 to 0.008830] | 0.003300 [0.001670 to 0.005510] | 0.010000 [0.002650 to 0.028000] | 0.010000 [0.002740 to 0.015000]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 120 | 0.002705 [0.000000 to 0.005470] | 0.001460 [0.000000 to 0.003000] | 0.012000 [0.002670 to 0.035000] | 0.006000 [0.002230 to 0.013000]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 120 | 0.000975 [0.000000 to 0.002670] | 0.001220 [0.000000 to 0.001840] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.001580] | 0.000000 [0.000000 to 0.001150] | 0.000000 [0.000000 to 0.001920] | 0.000000 [0.000000 to 0.001460]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 120 | 0.000000 [0.000000 to 0.000908] | 0.000000 [0.000000 to 0.000953] | 0.001540 [0.000000 to 0.003450] | 0.000000 [0.000000 to 0.001650]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 120 | 0.002885 [0.000760 to 0.005320] | 0.002070 [0.000000 to 0.003680] | 0.007155 [0.000000 to 0.036000] | 0.007850 [0.000000 to 0.028000]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 120 | 0.002915 [0.001090 to 0.004370] | 0.000450 [0.000000 to 0.002670] | 0.144565 [0.039110 to 0.447000] | 0.093000 [0.053410 to 0.163270]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 120 | 0.000702 [0.000000 to 0.003690] | 0.001570 [0.000000 to 0.002150] | 0.102525 [0.039880 to 0.291210] | 0.078900 [0.025190 to 0.134400]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 120 | 0.004735 [0.000280 to 0.013000] | 0.011430 [0.003910 to 0.017000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 120 | 0.000530 [0.000000 to 0.005520] | 0.000000 [0.000000 to 0.003730] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001140]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 120 | 0.003100 [0.000000 to 0.007000] | 0.006490 [0.000000 to 0.010660] | 0.000000 [0.000000 to 0.001420] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 120 | 0.001520 [0.000000 to 0.004710] | 0.002490 [0.000000 to 0.005030] | 0.004280 [0.001060 to 0.009270] | 0.004080 [0.000000 to 0.016790]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 120 | 0.001235 [0.000000 to 0.002480] | 0.000190 [0.000000 to 0.002720] | 0.046825 [0.015000 to 0.111210] | 0.024000 [0.007000 to 0.056110]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 120 | 0.000020 [0.000000 to 0.002480] | 0.000000 [0.000000 to 0.002260] | 0.034610 [0.011000 to 0.101210] | 0.016280 [0.006480 to 0.030630]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 120 | 0.009500 [0.000000 to 0.011000] | 0.006000 [0.000000 to 0.015000] | 0.001500 [0.000000 to 0.017000] | 0.002000 [0.000000 to 0.014000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 120 | 0.000000 [0.000000 to 0.007000] | 0.002000 [0.000000 to 0.011000] | 0.000500 [0.000000 to 0.019000] | 0.003000 [0.000000 to 0.012000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 120 | 0.000000 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.013000] | 0.000000 [0.000000 to 0.011000] | 0.006000 [0.000000 to 0.020000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 120 | 0.007000 [0.000000 to 0.040000] | 0.000000 [0.000000 to 0.019000] | 0.004500 [0.000000 to 0.028000] | 0.000000 [0.000000 to 0.014000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 120 | 0.008000 [0.000000 to 0.030000] | 0.000000 [0.000000 to 0.028000] | 0.018000 [0.000000 to 0.034000] | 0.009000 [0.000000 to 0.019000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 120: number analyzed (Participants) | 42 | 33 | 42 | 33
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 120 | 0.020000 [0.000000 to 0.050000] | 0.010000 [0.000000 to 0.040000] | 0.016500 [0.000000 to 0.040000] | 0.008000 [0.000000 to 0.023050]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Day 270 | 0.008790 [0.002970 to 0.019000] | 0.004355 [0.002620 to 0.011890] | 0.000000 [0.000000 to 0.002760] | 0.000411 [0.000000 to 0.002420]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Day 270 | 0.003410 [0.000000 to 0.006810] | 0.002170 [0.000355 to 0.004995] | 0.008760 [0.002360 to 0.020000] | 0.002605 [0.000010 to 0.008395]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Day 270 | 0.002890 [0.001110 to 0.005160] | 0.002720 [0.000059 to 0.005480] | 0.003960 [0.001120 to 0.026000] | 0.004575 [0.000000 to 0.012420]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.000980] | 0.000000 [0.000000 to 0.000505] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001930] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000635] | 0.000000 [0.000000 to 0.001570] | 0.000000 [0.000000 to 0.001150]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Day 270 | 0.001650 [0.000000 to 0.004170] | 0.000190 [0.000000 to 0.002215] | 0.003430 [0.000000 to 0.019000] | 0.008115 [0.000030 to 0.024475]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Day 270 | 0.001470 [0.000000 to 0.003600] | 0.000803 [0.000000 to 0.003250] | 0.099000 [0.036000 to 0.289000] | 0.069910 [0.027000 to 0.176500]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.002240] | 0.000798 [0.000000 to 0.002785] | 0.070000 [0.029000 to 0.258000] | 0.055015 [0.016265 to 0.128520]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Day 270 | 0.003230 [0.000000 to 0.009190] | 0.005735 [0.001130 to 0.013520] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.004920] | 0.000515 [0.000000 to 0.004630] | 0.000000 [0.000000 to 0.000055] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Day 270 | 0.001000 [0.000000 to 0.003470] | 0.002470 [0.000000 to 0.007075] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.001470]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.002800] | 0.000000 [0.000000 to 0.001245] | 0.003060 [0.000000 to 0.008450] | 0.003350 [0.000000 to 0.008815]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Day 270 | 0.000330 [0.000000 to 0.002550] | 0.000000 [0.000000 to 0.001390] | 0.022120 [0.002960 to 0.032080] | 0.007160 [0.002385 to 0.016904]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.003160] | 0.000000 [0.000000 to 0.002085] | 0.015270 [0.000620 to 0.033830] | 0.008945 [0.002924 to 0.027280]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.006000] | 0.001500 [0.000000 to 0.010500] | 0.000000 [0.000000 to 0.006000] | 0.001000 [0.000000 to 0.008500]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 39 | 31 | 39 | 32
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Day 270 | 0.000000 [0.000000 to 0.004000] | 0.000000 [0.000000 to 0.001000] | 0.000000 [0.000000 to 0.005000] | 0.000000 [0.000000 to 0.003500]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Day 270 | 0.000000 [0.000000 to 0.007000] | 0.000000 [0.000000 to 0.007500] | 0.000000 [0.000000 to 0.007460] | 0.000000 [0.000000 to 0.005500]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Day 270 | 0.000000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.005000] | 0.003000 [0.000000 to 0.029000] | 0.000000 [0.000000 to 0.015000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Day 270 | 0.019000 [0.000000 to 0.050000] | 0.000000 [0.000000 to 0.011500] | 0.026000 [0.006000 to 0.070000] | 0.004000 [0.000000 to 0.028500]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 270: number analyzed (Participants) | 39 | 32 | 39 | 32
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Day 270 | 0.009000 [0.000000 to 0.050000] | 0.000000 [0.000000 to 0.027000] | 0.015000 [0.004000 to 0.047000] | 0.006000 [0.000000 to 0.024500]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 1 | 0.006710 [0.001620 to 0.010000] | 0.000000 [0.000000 to 0.004370] | 0.000000 [0.000000 to 0.002310] | 0.000000 [0.000000 to 0.000870]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 1 | 0.002960 [0.000000 to 0.006980] | 0.001590 [0.000000 to 0.004050] | 0.000170 [0.000000 to 0.005020] | 0.002000 [0.000000 to 0.003420]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 1 | 0.003220 [0.000000 to 0.007550] | 0.000000 [0.000000 to 0.002285] | 0.002460 [0.000000 to 0.010000] | 0.001200 [0.000000 to 0.004260]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 1 | 0.000745 [0.000000 to 0.001700] | 0.000000 [0.000000 to 0.002180] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.001240] | 0.000000 [0.000000 to 0.001510] | 0.000000 [0.000000 to 0.001330] | 0.000000 [0.000000 to 0.000060]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 1 | 0.000000 [0.000000 to 0.001620] | 0.000000 [0.000000 to 0.000789] | 0.000000 [0.000000 to 0.000961] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 1 | 0.001110 [0.000000 to 0.004180] | 0.000920 [0.000000 to 0.002310] | 0.000000 [0.000000 to 0.015000] | 0.000000 [0.000000 to 0.007750]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 1 | 0.001430 [0.000240 to 0.002718] | 0.000170 [0.000000 to 0.002810] | 0.033910 [0.007790 to 0.061950] | 0.013000 [0.004000 to 0.038490]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 1 | 0.001058 [0.000000 to 0.003260] | 0.000522 [0.000000 to 0.002760] | 0.036130 [0.006450 to 0.126150] | 0.010120 [0.001030 to 0.040000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 1 | 0.003000 [0.000000 to 0.011820] | 0.003000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.001260] | 0.000000 [0.000000 to 0.001020]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 1 | 0.003000 [0.000000 to 0.006820] | 0.001000 [0.000000 to 0.005000] | 0.000000 [0.000000 to 0.000794] | 0.000000 [0.000000 to 0.001130]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 1 | 0.002000 [0.000000 to 0.011000] | 0.004000 [0.000000 to 0.012000] | 0.000000 [0.000000 to 0.001680] | 0.000000 [0.000000 to 0.001330]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 1 | 0.000190 [0.000000 to 0.002580] | 0.000746 [0.000000 to 0.002670] | 0.000000 [0.000000 to 0.006880] | 0.001300 [0.000000 to 0.005200]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.001802] | 0.000000 [0.000000 to 0.002430] | 0.003000 [0.000000 to 0.012095] | 0.003150 [0.000000 to 0.009260]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 1 | 0.000070 [0.000000 to 0.001880] | 0.000000 [0.000000 to 0.001900] | 0.003000 [0.000000 to 0.025100] | 0.003800 [0.000000 to 0.012000]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 1 | 0.000000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.010000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.010000] | 0.002000 [0.000000 to 0.015000] | 0.000000 [0.000000 to 0.007000] | 0.000000 [0.000000 to 0.009000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 1 | 0.000000 [0.000000 to 0.018000] | 0.006000 [0.000000 to 0.020000] | 0.001000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.010000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 1 | 0.000000 [0.000000 to 0.060000] | 0.020000 [0.000000 to 0.060000] | 0.000000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.003000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 1 | 0.000000 [0.000000 to 0.090000] | 0.010000 [0.000000 to 0.060000] | 0.006000 [0.000000 to 0.024000] | 0.004420 [0.000000 to 0.017000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 1: number analyzed (Participants) | 39 | 31 | 39 | 31
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 1 | 0.057000 [0.000000 to 0.100000] | 0.034000 [0.000000 to 0.140000] | 0.007000 [0.000000 to 0.031000] | 0.007000 [0.000000 to 0.017420]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 2 | 0.003744 [0.001870 to 0.009000] | 0.001200 [0.000000 to 0.003920] | 0.000000 [0.000000 to 0.001040] | 0.000000 [0.000000 to 0.001100]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 2 | 0.000613 [0.000000 to 0.004954] | 0.000860 [0.000000 to 0.002303] | 0.002100 [0.000786 to 0.004890] | 0.000042 [0.000000 to 0.002950]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 2 | 0.001490 [0.000000 to 0.003990] | 0.001510 [0.000050 to 0.005870] | 0.001700 [0.000000 to 0.005170] | 0.001340 [0.000000 to 0.005320]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.001820] | 0.000000 [0.000000 to 0.000948] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.000751] | 0.000000 [0.000000 to 0.000954] | 0.000000 [0.000000 to 0.000030] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 2 | 0.000000 [0.000000 to 0.002170] | 0.000000 [0.000000 to 0.000803] | 0.000000 [0.000000 to 0.000953] | 0.000000 [0.000000 to 0.001190]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 2 | 0.001190 [0.000045 to 0.001810] | 0.000120 [0.000000 to 0.002640] | 0.001720 [0.000000 to 0.006280] | 0.000000 [0.000000 to 0.002570]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.001950] | 0.000150 [0.000000 to 0.000948] | 0.025000 [0.008990 to 0.067240] | 0.007800 [0.002640 to 0.046410]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 2 | 0.000631 [0.000000 to 0.002210] | 0.001390 [0.000000 to 0.002410] | 0.015650 [0.002880 to 0.054000] | 0.012220 [0.003480 to 0.028820]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 2 | 0.001000 [0.000000 to 0.005000] | 0.000380 [0.000000 to 0.003510] | 0.000000 [0.000000 to 0.000835] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 2 | 0.000760 [0.000000 to 0.006670] | 0.000000 [0.000000 to 0.003070] | 0.000000 [0.000000 to 0.000852] | 0.000000 [0.000000 to 0.001130]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 2 | 0.002000 [0.000000 to 0.008760] | 0.005000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.000940] | 0.000000 [0.000000 to 0.000947]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 2 | 0.000320 [0.000000 to 0.002130] | 0.000588 [0.000000 to 0.002100] | 0.000670 [0.000000 to 0.001940] | 0.000000 [0.000000 to 0.002020]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 2 | 0.000180 [0.000000 to 0.001130] | 0.000578 [0.000000 to 0.001680] | 0.004920 [0.002000 to 0.007370] | 0.003380 [0.000130 to 0.007030]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 2 | 0.000621 [0.000000 to 0.001449] | 0.000017 [0.000000 to 0.001550] | 0.004580 [0.000000 to 0.009150] | 0.001140 [0.000000 to 0.007210]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.004000] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.005000] | 0.000000 [0.000000 to 0.007000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 2 | 0.000000 [0.000000 to 0.002000] | 0.000000 [0.000000 to 0.002000] | 0.000000 [0.000000 to 0.003000] | 0.000000 [0.000000 to 0.006000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 2 | 0.000000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.016000] | 0.000000 [0.000000 to 0.005360] | 0.000000 [0.000000 to 0.009000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 2 | 0.000000 [0.000000 to 0.049000] | 0.000000 [0.000000 to 0.022000] | 0.000000 [0.000000 to 0.004640] | 0.000000 [0.000000 to 0.000000]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 2 | 0.011000 [0.000000 to 0.050000] | 0.006000 [0.000000 to 0.060000] | 0.008310 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.014000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 2: number analyzed (Participants) | 31 | 25 | 31 | 25
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 2 | 0.044000 [0.001000 to 0.100000] | 0.018000 [0.000000 to 0.110000] | 0.004000 [0.000000 to 0.020000] | 0.000000 [0.000000 to 0.014300]
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2+TNFa+, DENV-2, NS1-2, Year 3 | 0.003110 [0.000000 to 0.008297] | 0.001934 [0.000180 to 0.004290] | 0.000000 [0.000000 to 0.001070] | 0.000000 [0.000000 to 0.001460]
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2+TNFa+, DENV-2, NS3-2, Year 3 | 0.000645 [0.000000 to 0.007000] | 0.000760 [0.000000 to 0.006250] | 0.000060 [0.000000 to 0.003050] | 0.001830 [0.000000 to 0.004090]
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2+TNFa+, DENV-2, NS5-2, Year 3 | 0.002612 [0.000000 to 0.007300] | 0.002510 [0.000000 to 0.003800] | 0.001420 [0.000000 to 0.006330] | 0.000000 [0.000000 to 0.002690]
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2+TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.000831] | 0.000000 [0.000000 to 0.001180] | 0.000000 [0.000000 to 0.000000] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2+TNFa-, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.001240] | 0.000778 [0.000000 to 0.001670] | 0.000000 [0.000000 to 0.000811] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2+TNFa-, DENV-2, NS5-2, Year 3 | 0.000686 [0.000000 to 0.002770] | 0.000000 [0.000000 to 0.002070] | 0.000000 [0.000000 to 0.001290] | 0.000000 [0.000000 to 0.000000]
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2-TNFa+, DENV-2, NS1-2, Year 3 | 0.000070 [0.000000 to 0.002070] | 0.000557 [0.000000 to 0.001940] | 0.000000 [0.000000 to 0.003040] | 0.000000 [0.000000 to 0.002560]
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2-TNFa+, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.001660] | 0.000000 [0.000000 to 0.001574] | 0.012470 [0.002000 to 0.023163] | 0.004220 [0.000210 to 0.014900]
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2-TNFa+, DENV-2, NS5-2, Year 3 | 0.000000 [0.000000 to 0.001580] | 0.001050 [0.000000 to 0.002364] | 0.007735 [0.001000 to 0.053360] | 0.007770 [0.000832 to 0.029000]
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2+TNFa+, DENV-2, NS1-2, Year 3 | 0.001740 [0.000000 to 0.005570] | 0.001650 [0.000000 to 0.004000] | 0.000000 [0.000000 to 0.000873] | 0.000000 [0.000000 to 0.000930]
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2+TNFa+, DENV-2, NS3-2, Year 3 | 0.000880 [0.000000 to 0.002680] | 0.001000 [0.000000 to 0.003810] | 0.000000 [0.000000 to 0.000750] | 0.000000 [0.000000 to 0.001890]
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2+TNFa+, DENV-2, NS5-2, Year 3 | 0.001500 [0.000000 to 0.008170] | 0.002170 [0.000000 to 0.006000] | 0.000000 [0.000000 to 0.001230] | 0.000000 [0.000000 to 0.000150]
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2-TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.000702] | 0.000864 [0.000000 to 0.002005] | 0.000000 [0.000000 to 0.001820] | 0.000090 [0.000000 to 0.002680]
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2-TNFa-, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.001637] | 0.000000 [0.000000 to 0.001310] | 0.002707 [0.000000 to 0.006560] | 0.002320 [0.000000 to 0.006260]
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg+IL2-TNFa-, DENV-2, NS5-2, Year 3 | 0.000523 [0.000000 to 0.001820] | 0.000010 [0.000000 to 0.001560] | 0.002955 [0.000000 to 0.011250] | 0.001070 [0.000000 to 0.006670]
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2+TNFa-, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.006000] | 0.000000 [0.000000 to 0.009000] | 0.000040 [0.000000 to 0.005000] | 0.000000 [0.000000 to 0.003000]
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2+TNFa-, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.010000] | 0.003000 [0.000000 to 0.009000] | 0.000000 [0.000000 to 0.004830] | 0.000000 [0.000000 to 0.010000]
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2+TNFa-, DENV-2, NS5-2, Year 3 | 0.000500 [0.000000 to 0.015000] | 0.004000 [0.000000 to 0.013000] | 0.000500 [0.000000 to 0.007000] | 0.000000 [0.000000 to 0.006000]
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2-TNFa+, DENV-2, NS1-2, Year 3 | 0.000000 [0.000000 to 0.030000] | 0.000000 [0.000000 to 0.010000] | 0.000000 [0.000000 to 0.004000] | 0.000000 [0.000000 to 0.011710]
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2-TNFa+, DENV-2, NS3-2, Year 3 | 0.000000 [0.000000 to 0.011000] | 0.000000 [0.000000 to 0.012000] | 0.004000 [0.000000 to 0.014000] | 0.001270 [0.000000 to 0.026000]
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 3: number analyzed (Participants) | 38 | 31 | 38 | 31
  IFNg-IL2-TNFa+, DENV-2, NS5-2, Year 3 | 0.023000 [0.000000 to 0.060000] | 0.016000 [0.000000 to 0.070000] | 0.003000 [0.000000 to 0.016000] | 0.008000 [0.000000 to 0.018000]

14. Secondary Outcome: Geometric Mean Titers (GMT) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 1 Month Post First Vaccination, Pre Second Vaccination, and 1, 6 Months Post Second Vaccination and Then Annually Up to 3 Years
Description: GMT of neutralizing antibodies was measured by microneutralization test (MTN). The dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: 1 month post first vaccination (Day 30); pre second vaccination (Day 90); 1 and 6 months post second vaccination (Days 120 and 270); annually up to 3 years (Years 1, 2 and 3)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 195
titer
  DENV-1, Day 30: number analyzed (Participants) | 185
  DENV-1, Day 30 | 402.3 [287.5 to 562.9]
  DENV-2, Day 30: number analyzed (Participants) | 185
  DENV-2, Day 30 | 5482.2 [4626.4 to 6496.3]
  DENV-3, Day 30: number analyzed (Participants) | 185
  DENV-3, Day 30 | 436.1 [326.9 to 581.7]
  DENV-4, Day 30: number analyzed (Participants) | 185
  DENV-4, Day 30 | 253.9 [182.6 to 353.1]
  DENV-1, Day 90 | 271.7 [193.9 to 380.7]
  DENV-2, Day 90 | 2736.3 [2295.1 to 3262.5]
  DENV-3, Day 90 | 218.7 [162.0 to 295.2]
  DENV-4, Day 90 | 177.4 [129.6 to 242.8]
  DENV-1, Day 120: number analyzed (Participants) | 182
  DENV-1, Day 120 | 550.6 [408.0 to 743.1]
  DENV-2, Day 120: number analyzed (Participants) | 182
  DENV-2, Day 120 | 2808.2 [2395.0 to 3292.8]
  DENV-3, Day 120: number analyzed (Participants) | 182
  DENV-3, Day 120 | 404.2 [312.6 to 522.7]
  DENV-4, Day 120: number analyzed (Participants) | 182
  DENV-4, Day 120 | 427.1 [335.4 to 543.8]
  DENV-1, Day 270: number analyzed (Participants) | 187
  DENV-1, Day 270 | 343.3 [249.8 to 471.6]
  DENV-2, Day 270: number analyzed (Participants) | 187
  DENV-2, Day 270 | 1729.9 [1435.7 to 2084.4]
  DENV-3, Day 270: number analyzed (Participants) | 187
  DENV-3, Day 270 | 203.8 [153.5 to 270.7]
  DENV-4, Day 270: number analyzed (Participants) | 187
  DENV-4, Day 270 | 186.6 [141.6 to 246.0]
  DENV-1, Year 1: number analyzed (Participants) | 192
  DENV-1, Year 1 | 243.8 [176.4 to 337.0]
  DENV-2, Year 1: number analyzed (Participants) | 192
  DENV-2, Year 1 | 896.2 [729.9 to 1100.5]
  DENV-3, Year 1: number analyzed (Participants) | 192
  DENV-3, Year 1 | 148.6 [111.6 to 197.7]
  DENV-4, Year 1: number analyzed (Participants) | 192
  DENV-4, Year 1 | 142.4 [108.8 to 186.3]
  DENV-1, Year 2: number analyzed (Participants) | 154
  DENV-1, Year 2 | 290.8 [200.8 to 421.1]
  DENV-2, Year 2: number analyzed (Participants) | 154
  DENV-2, Year 2 | 724.7 [564.2 to 930.8]
  DENV-3, Year 2: number analyzed (Participants) | 154
  DENV-3, Year 2 | 172.7 [120.6 to 247.1]
  DENV-4, Year 2: number analyzed (Participants) | 154
  DENV-4, Year 2 | 157.7 [114.0 to 218.0]
  DENV-1, Year 3: number analyzed (Participants) | 180
  DENV-1, Year 3 | 178.7 [127.3 to 250.8]
  DENV-2, Year 3: number analyzed (Participants) | 180
  DENV-2, Year 3 | 546.4 [435.2 to 686.0]
  DENV-3, Year 3: number analyzed (Participants) | 180
  DENV-3, Year 3 | 125.2 [92.8 to 169.0]
  DENV-4, Year 3: number analyzed (Participants) | 180
  DENV-4, Year 3 | 91.6 [69.4 to 120.7]

15. Secondary Outcome: Percentage of Participants Seropositive for Each of the 4 Dengue Serotypes at 1 Month Post First Vaccination, Pre-second Vaccination, and 1, 6 Months Post Second Vaccination and Then Annually up to 3 Years
Description: Seropositive was defined as a reciprocal neutralizing titer ≥10. The dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: as for outcome 14
Population: PPS included all participants from the FAS who have no major protocol violations. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 195
percentage of participants
  DENV-1, Day 30: number analyzed (Participants) | 185
  DENV-1, Day 30 | 96.8 [93.1 to 98.8]
  DENV-2, Day 30: number analyzed (Participants) | 185
  DENV-2, Day 30 | 99.5 [97.0 to 100.0]
  DENV-3, Day 30: number analyzed (Participants) | 185
  DENV-3, Day 30 | 99.5 [97.0 to 100.0]
  DENV-4, Day 30: number analyzed (Participants) | 185
  DENV-4, Day 30 | 93.0 [88.3 to 96.2]
  DENV-1, Day 90 | 90.8 [85.8 to 94.4]
  DENV-2, Day 90 | 99.5 [97.2 to 100.0]
  DENV-3, Day 90 | 94.4 [90.1 to 97.2]
  DENV-4, Day 90 | 91.8 [87.0 to 95.2]
  DENV-1, Day 120: number analyzed (Participants) | 182
  DENV-1, Day 120 | 99.5 [97.0 to 100.0]
  DENV-2, Day 120: number analyzed (Participants) | 182
  DENV-2, Day 120 | 100.0 [98.0 to 100.0]
  DENV-3, Day 120: number analyzed (Participants) | 182
  DENV-3, Day 120 | 100.0 [98.0 to 100.0]
  DENV-4, Day 120: number analyzed (Participants) | 182
  DENV-4, Day 120 | 100.0 [98.0 to 100.0]
  DENV-1, Day 270: number analyzed (Participants) | 187
  DENV-1, Day 270 | 96.8 [93.1 to 98.8]
  DENV-2, Day 270: number analyzed (Participants) | 187
  DENV-2, Day 270 | 100.0 [98.0 to 100.0]
  DENV-3, Day 270: number analyzed (Participants) | 187
  DENV-3, Day 270 | 97.9 [94.6 to 99.4]
  DENV-4, Day 270: number analyzed (Participants) | 187
  DENV-4, Day 270 | 96.8 [93.1 to 98.8]
  DENV-1, Year 1: number analyzed (Participants) | 192
  DENV-1, Year 1 | 91.1 [86.2 to 94.8]
  DENV-2, Year 1: number analyzed (Participants) | 192
  DENV-2, Year 1 | 100.0 [98.1 to 100.0]
  DENV-3, Year 1: number analyzed (Participants) | 192
  DENV-3, Year 1 | 93.8 [89.3 to 96.7]
  DENV-4, Year 1: number analyzed (Participants) | 192
  DENV-4, Year 1 | 96.4 [92.6 to 98.5]
  DENV-1, Year 2: number analyzed (Participants) | 154
  DENV-1, Year 2 | 93.5 [88.4 to 96.8]
  DENV-2, Year 2: number analyzed (Participants) | 154
  DENV-2, Year 2 | 100.0 [97.6 to 100.0]
  DENV-3, Year 2: number analyzed (Participants) | 154
  DENV-3, Year 2 | 89.6 [83.7 to 93.9]
  DENV-4, Year 2: number analyzed (Participants) | 154
  DENV-4, Year 2 | 95.5 [90.9 to 98.2]
  DENV-1, Year 3: number analyzed (Participants) | 180
  DENV-1, Year 3 | 84.4 [78.3 to 89.4]
  DENV-2, Year 3: number analyzed (Participants) | 180
  DENV-2, Year 3 | 100.0 [98.0 to 100.0]
  DENV-3, Year 3: number analyzed (Participants) | 180
  DENV-3, Year 3 | 86.7 [80.8 to 91.3]
  DENV-4, Year 3: number analyzed (Participants) | 180
  DENV-4, Year 3 | 86.1 [80.2 to 90.8]

16. Secondary Outcome: Percentage of Participants Seropositive for Multiple Dengue Serotypes at 1 Month Post First Vaccination, Pre Second Vaccination, 1, 6 Months Post Second Vaccination and Annually up to 3 Years
Description: Seropositive was defined as a reciprocal neutralizing titer ≥10. The dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Seropositive for multiple dengue serotypes were summarized in the following categories: tetravalent and at least trivalent.
Time Frame: as for outcome 14
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 195
percentage of participants
  Tetravalent, Day 30: number analyzed (Participants) | 185
  Tetravalent, Day 30 | 90.8 [85.7 to 94.6]
  At Least Trivalent, Day 30: number analyzed (Participants) | 185
  At Least Trivalent, Day 30 | 98.4 [95.3 to 99.7]
  Tetravalent, Day 90 | 83.6 [77.6 to 88.5]
  At Least Trivalent, Day 90 | 95.4 [91.4 to 97.9]
  Tetravalent, Day 120: number analyzed (Participants) | 182
  Tetravalent, Day 120 | 99.5 [97.0 to 100.0]
  At Least Trivalent, Day 120: number analyzed (Participants) | 182
  At Least Trivalent, Day 120 | 100.0 [98.0 to 100.0]
  Tetravalent, Day 270: number analyzed (Participants) | 187
  Tetravalent, Day 270 | 93.0 [88.4 to 96.2]
  At Least Trivalent, Day 270: number analyzed (Participants) | 187
  At Least Trivalent, Day 270 | 98.4 [95.4 to 99.7]
  Tetravalent, Year 1: number analyzed (Participants) | 192
  Tetravalent, Year 1 | 87.5 [82.0 to 91.8]
  At Least Trivalent, Year 1: number analyzed (Participants) | 192
  At Least Trivalent, Year 1 | 95.3 [91.3 to 97.8]
  Tetravalent, Year 2: number analyzed (Participants) | 154
  Tetravalent, Year 2 | 86.4 [79.9 to 91.4]
  At Least Trivalent, Year 2: number analyzed (Participants) | 154
  At Least Trivalent, Year 2 | 93.5 [88.4 to 96.8]
  Tetravalent, Year 3: number analyzed (Participants) | 180
  Tetravalent, Year 3 | 76.7 [69.8 to 82.6]
  At Least Trivalent, Year 3: number analyzed (Participants) | 180
  At Least Trivalent, Year 3 | 87.2 [81.4 to 91.7]

17. Secondary Outcome: Percentage of Participants Experiencing Unsolicited Adverse Events (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration.
Time Frame: Up to 28 days (day of vaccination + 27 days) after administration of each vaccine dose on Day 1 [Month 0] and Day 90 [Month 3]
Population: Safety Set included all enrolled participants who received at least 1 dose of TDV. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 200
percentage of participants
  After First Vaccination | 26.5
  After Second Vaccination: number analyzed (Participants) | 198
  After Second Vaccination | 25.3

18. Secondary Outcome: Percentage of Participants With Medically Attended AEs (MAAEs)
Description: MAAEs were defined as AEs leading to a medical visit to or by a healthcare professional, including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: From first vaccination (Day 1) up to 6 months post second vaccination (Day 270)
Population: Safety Set included all enrolled participants who received at least 1 dose of TDV.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 200
percentage of participants | 50.5

19. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A SAE was defined as any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From first vaccination (Day 1) up to end of study (Approximately 3 years)
Population: Safety Set included all enrolled participants who received at least 1 dose of TDV.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 200
percentage of participants | 5.5

20. Secondary Outcome: Percentage of Participants With Virologically Confirmed Dengue
Description: Participants with febrile illness defined as fever ≥38°C on any 2 of 3 consecutive days were evaluated for dengue. Virologically confirmed dengue was defined as febrile illness with a positive serotype-specific RT-PCR (i.e. positive dengue detection RT-PCR).
Time Frame: From first vaccination (Day 1) up to 6 months post second vaccination (Day 270)
Population: Safety Set included all enrolled participants who received at least 1 dose of TDV.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
Number analyzed (Participants) | 200
percentage of participants | 6.0

ADVERSE EVENTS:
Time Frame: All-cause mortality and Serious adverse events: From first vaccination (Day 1) up to end of study (Approximately 3 years); Non-serious adverse events: Up to 28 days (day of vaccination + 27 days) after administration of each vaccine dose on Day 1 [Month 0] and Day 90 [Month 3]
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Tetravalent Dengue Vaccine (TDV) 0.5 mL
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 11/200
Other Adverse Events (participants affected / at risk) | 66/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tetravalent Dengue Vaccine (TDV) 0.5 mL (N=200)
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Typhoid fever (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Dengue fever (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Systemic viral infection (Infections and infestations) | 1
Febrile convulsion (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Victim of sexual abuse (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tetravalent Dengue Vaccine (TDV) 0.5 mL (N=200)
Nasopharyngitis (Infections and infestations) | 29
Upper respiratory tract infection (Infections and infestations) | 20
Gastroenteritis (Infections and infestations) | 12
Systemic viral infection (Infections and infestations) | 9
Pneumonia (Infections and infestations) | 8
Conjunctivitis (Infections and infestations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT02948829/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT02948829/SAP_001.pdf